CLINICAL TRIAL: NCT02201433
Title: Study on the Treatment of Children and Their Families in Services Related to Early Childhood Morvan Hospital Qualitative Study
Brief Title: Study on the Treatment of Children and Their Families in Services Related to Early Childhood
Acronym: PERAM-QUAL
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: PERAM-QUAL
Record Dates: First submitted 2014-07-09; First posted 2014-07-28 (Estimated); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Fathers; Premature Birth
Keywords: breastfeeding; fathers; preterm newborns; partner influence
MeSH Terms: conditions — Premature Birth; Breast Feeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- medical staff and member of an association: members of medical staff and member of an association of parents of premature infants.
  This cohort is necessary to build protocol interview for part 2 of the study
- fathers: fathers of preterm newborns
- fathers or médical staff: This cohort is build for data validation. We will include fathers who have experienced this situation. Caregivers of NICU who are not participating in the first part

SUMMARY:
Breastfeeding is recommended for preterm infants. Development of breastfeeding is an important issue, requiring the involvement of medical and paramedical staff in neonatal units. There are few data concerning the fathers of preterm infants. However, the role of the father is identified in the literature as a key factor in the initiation and continuation of breastfeeding. In our neonatal unit care, reasons for breastfeeding high rates are not identified but may be related to the father being in close and constant contact with the medical and paramedical staff. In fact, fathers are often first in contact with caregivers. They can be invested in the implementation of nursing care, skin to skin, as well as being asked to support the development of their child in the service and at home.

The aims of this study are to:

* Analyze the beliefs, social representations and the experience of the fathers of premature infants hospitalized in intensive care unit concerning breastfeeding.
* Analyze the factors facilitating and inhibiting the initiation and continuation of breastfeeding.
* Consider strategies of care and support that can be used for the families of premature infants and of children born at term.
* Explore the expectations of medical staff with regards to the management of children and families, their practices, identify the role attributed to the father.
* Initiate and facilitate reflexivity of medical and paramedical staff about their respective practices

DETAILED DESCRIPTION:
The study will be conducted in three phases according to the methodology of qualitative research:

* The first for the preparation of interview guides and observation grids through the inclusion of 20 participants: caregivers and members of associations of preterm parents,
* The second part: maintenance by the inclusion of 40 fathers of children born preterm before 37 weeks and their partner if she wants.
* The third part will, as in any qualitative analysis, data validation with the inclusion of 20 participants: fathers who experienced this situation in the context of care and caregivers close to neonatal intensive unit care (NICU) are participants in the first phase.

interview methods:

* 1 exploratory interview two hours on average with each part 1 and part 3 participants.
* 3-5 interviews per part 2 participant. Interviews are conduct with guideline constructed during the first part of the study. Interview will be conducted by a nurse and /or a psychologist

Data analysis:

Full transcript of the interviews. Partial treatment during the study to enrich the interview guide until data saturation. All data will be treated differently: Software-aided thematic treatment (NVivo) and textual processing with cross medical data and socio-demographic variables (Alceste).

Data Validation :

Part 3 of the study external validation. Literature validation

ELIGIBILITY:
PART 1

Inclusion Criteria:

* Member of Association of Parents of premature children major (born before 37 weeks)
* Medical staff (doctors, nurses, pediatric nurses, social worker, ...) working in the NICU of the study.
* Signing of free and informed consent

PART 2

Inclusion Criteria:

* major fathers of child born before 37 weeks who survived to the early neonatal period (7days),
* French mother tongue,
* Residing in the geographical area of Brest
* Signing of free and informed consent
* Inclusion between Day 7 and Day 30 after the birth of their child

PART 3

Inclusion Criteria:

* fathers who have experienced child born premature
* caregivers of NICU

PART 1, 2 and 3 exclusion criteria:

* Person whose refuse to participate
* Persons unable to consent
* Persons whose monitoring is impossible
* minor

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Part 1: caregivers and members of associations of preterm parents Part 2: fathers of preterm newborns, hospitalized in a neonatal intensive care unit Part 3: fathers who have experienced premature and caregivers of NICU who not participating in the first part
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Interviews | Day 7
  PERAM QUAL is a qualitative study, in accordance with the methodology of qualitative study, it is not possible to establish a quantitative criterion of judgment.
  Full transcript of the interviews should permit the identification of factors that promote breastfeeding.

CONTACTS AND LOCATIONS:
Overall Officials: HELENE DENOUAL, Principal Investigator — University Hospital, Brest
Locations (2):
- France (2):
  - CHRU de Brest, Brest
  - CH du Mans, Le Mans